CLINICAL TRIAL: NCT03342859
Title: An Open-label, Parallel Group, Multi-center Study to Investigate Pharmacodynamic Effects After Daily Administration of Vilaprisan or Ulipristal Acetate for 8-12 Weeks in Patients With Uterine Fibroids for Whom Surgery (Hysterectomy or Myomectomy) is Planned
Brief Title: Mode of Action Study of Vilaprisan and Ulipristal Acetate in Patients With Uterine Fibroids for Whom Surgery is Planned
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to findings in the preclinical carcinogenicity studies for vilaprisan (BAY1002670)
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15791; 2017-000468-13 (EudraCT Number)
Record Dates: First submitted 2017-10-26; First posted 2017-11-17 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Leiomyoma
Keywords: Uterine fibroids; Bleeding reduction; Vilaprisan; Mode of action; Hysterectomy; Myomectomy; Pharmacodynamic
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan; ulipristal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vilaprisan group (Experimental): Vilaprisan 2 mg oral daily over 8-12 weeks
  Interventions: Drug: Vilaprisan, BAY1002670
- Ulipristal group (Active Comparator): Ulipristal 5 mg oral daily over 8-12 weeks
  Interventions: Drug: Ulipristal
- Control group (No Intervention): Patients undergoing surgery without any prior treatment, as control group

INTERVENTIONS:
Drug: Vilaprisan, BAY1002670 — Daily single oral doses of 2 mg vilaprisan over 8-12 weeks
  Arms: Vilaprisan group
Drug: Ulipristal — Daily single oral doses of 5 mg ulipristal over 8-12 weeks
  Arms: Ulipristal group

SUMMARY:
To investigate the clinical effects of vilaprisan and ulipristal acetate at molecular and cellular level on uterine and fibroid tissue taken from patients (after surgery / biopsy)

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older and premenopausal (based on gynecological history i.e. still menstruating; no significant estrogen deficiency symptoms)
* Diagnosis of uterine fibroids documented by ultrasound and relevant symptoms reported by the patient (e.g. heavy menstrual bleeding, pelvic pressure)
* Patients for whom surgery (hysterectomy or myomectomy) for the treatment of symptomatic uterine fibroids is planned
* Patients who are otherwise healthy as shown by medical history, physical and gynecological examinations, and laboratory test results

Exclusion Criteria:

* Contraindications for the progesterone receptor modulators (PRM) vilaprisan or ulipristal acetate
* Use of medication that might interfere with the conduct of the study or the interpretation of the results (e.g. continuing use of hormonal contraceptives, tranexamic acid or other treatments for heavy menstrual bleeding, progesterone receptor modulators, gonadotropin-releasing hormone agonist, anticoagulants, moderate and strong CYP3A4 inducers and moderate and strong CYP3A4 inhibitors within a defined time period before treatment starts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
The expression level of biomarker for glandular and stromal cell proliferation (Ki-67) in the endometrium of the same patient before treatment and when treated with VPR (vilaprisan) prior to surgery | From pre-treatment biopsy to post-treatment biopsy_ Up to 20 weeks
  Pre-treatment biopsy: The endometrial biopsy will be performed between Day 6 to 13 of the menstrual cycle that occurs after the screening visit and before treatment commences. Post-treatment biopsy as second endometrial biopsy is taken (if possible within 24 hours) after end of VPR treatment.
The expression level of biomarker for myoma cell proliferation (Ki-67) in fibroid tissue of patients not treated with PRM (progesterone receptor modulator )and those who have been treated with VPR prior to surgery | After maximum 12 weeks of treatment
  Fibroid tissue sample will be collected from the uterus following surgery (if possible within 24 hours) after end of VPR treatment
The expression level of biomarkers for apoptotic regulation in the endometrium (BCL-2 (B-cell lymphoma 2), caspase 3) of the same patient before treatment and when treated with VPR prior to surgery | From pre-treatment biopsy to post-treatment biopsy_ Up to 20 weeks
  Pre-treatment biopsy: The endometrial biopsy will be performed between Day 6 to 13 of the menstrual cycle that occurs after the screening visit and before treatment commences. Post-treatment biopsy as second endometrial biopsy is taken (if possible within 24 hours) after end of VPR treatment
The expression level of biomarkers for apoptotic regulation in fibroid tissue (BCL-2, caspase 3) of patients not treated with PRM and those who have been treated with VPR prior to surgery | After maximum 12 weeks of treatment
  Fibroid tissue sample will be collected from the uterus following surgery (if possible within 24 hours) after end of VPR treatment
The expression level of nuclear hormone receptors in the endometrium (progesterone receptor (PR), PR-B, estrogen receptor (ER), androgen receptor (AR)) of the same patient before treatment and when treated with VPR prior to surgery | From pre-treatment biopsy to post-treatment biopsy_ Up to 20 weeks
  Pre-treatment biopsy: The endometrial biopsy will be performed between Day 6 to 13 of the menstrual cycle that occurs after the screening visit and before treatment commences. Post-treatment biopsy as second endometrial biopsy is taken (if possible within 24 hours) after end of VPR treatment

SECONDARY OUTCOMES:
The expression levels of biomarkers (Ki-67, caspase 3 and BCL-2) in the endometrium of the same patient before treatment and when treated with UPA prior to surgery | From pre-treatment biopsy to post-treatment biopsy_ Up to 20 weeks
  Pre-treatment biopsy: The endometrial biopsy will be performed between Day 6 to 13 of the menstrual cycle that occurs after the screening visit and before treatment commences. Post-treatment biopsy as second endometrial biopsy is taken (if possible within 24 hours) after end of treatment. Fibroid tissue sample will be collected from the uterus following surgery (if possible within 24 hours) after end of treatment
The expression levels of biomarkers (Ki-67, caspase 3 and BCL-2) in fibriod tissue of patients not treated with PRM and those who have been treated with UPA prior to surgery | After maximum 12 weeks of treatment
  Fibroid tissue sample will be collected from the uterus following surgery (if possible within 24 hours) after end of VPR treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Edinburgh Royal Infirmary/ NHS Lothian, Edinburgh, United Kingdom

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/